CLINICAL TRIAL: NCT02427711
Title: Reduced Total Blood Loss and Blood Transfusion in Non-Septic Revision Knee Arthroplasty Using a Bipolar Sealer - A Prospective Cohort Study With Retrospective Controls
Brief Title: Reduced Total Blood Loss and Blood Transfusion in Non-Septic Revision Knee Arthroplasty Using a Bipolar Sealer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christian Skovgaard Nielsen, MD, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HVH-2013-037
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-04

CONDITIONS: Total Blood Loss
Keywords: Reduction of blood loss for revisions of knee arthroplasty; blood transfusions; Readmission; Bipolar sealer
MeSH Terms: conditions — Exsanguination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipolar sealer (Active Comparator): Prospective use of bipolar sealer for skin and knee capsule incision revisions of non-septic knee arthroplasty.
  Interventions: Device: Bipolar sealer
- Scalpel (Placebo Comparator): Conventional surgical incision with scalpel - data extracted from a retrospective group.
  Interventions: Device: Bipolar sealer

INTERVENTIONS:
Device: Bipolar sealer — Prospective trial with Aquamantys for surgical skin and capsula incision w a retrospective control group using a conventional scalpel skin and capsula incision.
  Other Names: Aquamantys

SUMMARY:
To investigate if the use of a bipolar sealer for skin and capsula incision results in decreased total blood loss and/or less blood transfusion in non-septic knee arthroplasty.

DETAILED DESCRIPTION:
In patients undergoing primary total knee arthroplasty, perioperative anemia is highly prevalent. In a systematic review, preoperative anemia was found in 24 +/- 9% and postoperative anemia in 51% +/- 10%. Perioperative anemia was associated with a blood transfusion rate of 45 +/- 25%, postoperative infections, poorer physical functioning and recovery, and increased length of hospital stay (LOS) and mortality. Although the best transfusion trigger in elective patients remains unknown, restrictive transfusion protocols are recommended and avoidance of blood transfusion if possible.

The only non-systemic modality capable of reducing blood loss before it occurs is a bipolar sealer (Aquamantys). By pre-incisional treatment of the soft tissue, bleeding (and potentially total blood loss and transfusion) is reduced without tissue charring.

Previously studies on the use of Aquamantys in primary knee arthroplasty have had various outcomes, the most recent being negative while the former 3 were positive regarding reduction in blood loss, drop in hgb and transfusions. No published date exist on potential outcomes in revision knee arthroplasty where blood loss and transfusion needs exceeds that of primary total knee arthroplasty by far. Aquamantys hence would theoretically benefit the most in a revision setting without the use of a tourniquet - and would be an interesting modality in modern contemporary fast-track revision if shown effective despite/on top of the use of additional blood saving modalities. The present study is therefore motivated by investigating this aspect.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Non septic knee-arthroplasty revision.
* Musk speak and understand Danish

Exclusion Criteria:

* Age below 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | 2nd postoperative morning

SECONDARY OUTCOMES:
Blood loss | 1st. postoperative morning
Blood transfusion | while hospitalized expected 5 days.
Readmission | 90 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark